CLINICAL TRIAL: NCT05469581
Title: Efficiency of Preventive Interventions in Community Nursing to Improve Medication Adherence in Vulnerable Elderly"
Brief Title: "Efficiency of Preventive Interventions in Community Nursing to Improve Medication Adherence in Vulnerable Elderly"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Martina Horvat (Other)
Responsible Party: Sponsor-Investigator, Martina Horvat, RN, community nursing specialist, PhD student/candidat, University Maribor
Organization: University Maribor (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 39641
Record Dates: First submitted 2022-07-03; First posted 2022-07-21 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Noncommunicable Diseases; Vulnerable Elderly
Keywords: Adherence; Medication; Preventive Interventions; Community Nursing; Vulnerable Elderly
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to two groups: experimental and control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Interventions to be administered:
  A set of preventive interventions to improve adherence in vulnerable elderly people (We will not administer any medications in the research):
  * reviewing the list of medications, delivery of an ordered list of medications and checking medication regimen understanding;
  * delivering a leaflet on the correct/safe taking of medication, discussion, explanation, and verification of understanding of the content;
  * a counseling about the importance of adherence;
  * handing over the medication dispenser (if the elderly person does not have one yet),
  * delivering of a personal medication card, which shows the timeline of taking prescribed medication.
  Interventions: Other: A set of preventive interventions to improve adherence in vulnerable elderly people
- Control group (No Intervention): Interventions to be administered:
  - review of the list of medication, delivery of an ordered list of medication, and counseling

INTERVENTIONS:
Other: A set of preventive interventions to improve adherence in vulnerable elderly people — * reviewing the list of medications, delivery of an ordered list of medications, and checking medication regimen understanding;
  * delivering a leaflet on the correct/safe taking of medications, discussion, explanation, and verification of understanding of the content;
  * a counseling about the importance of adherence;
  * handing over the medication dispenser (if the elderly person does not have one yet),
  * delivering of a personal medication card, which shows the timeline of taking prescribed medication.
  Arms: Intervention group

SUMMARY:
The purpose of the study is to design and investigate the effectiveness of a set of preventive interventions by community nurses in outpatient care in treating vulnerable elderly people to improve the extent to which they follow the agreed recommendations of a doctor or pharmacist regarding taking medication.

DETAILED DESCRIPTION:
We will conduct a randomized controlled trial to determine the effectiveness of preventive interventions to improve adherence in vulnerable elderly people.

The randomized controlled trial will include: vulnerable people over 65 years of age with preserved cognitive abilities who are receiving at least one medication for any medical condition and are being treated by an outpatient service; they live in their home environment, which in the first phase will show vulnerability and, at the same time, initial suboptimal adherence.

We will inform the subjects verbally and in writing about the course, purpose, and goals of the study and obtain their written consent for inclusion in the study. They will then be randomly assigned to two groups: experimental and control.

In the case of the experimental group, we will carry out a set of preventive interventions to support the improvement of medication adherence. The control group will receive regular nursing care from community nurses, to which we will add the so-called distractor.

We will determine the effectiveness of preventive interventions based on changes in self-efficacy and adherent behavior.

Data on adherence behavior and self-efficacy will be collected at the beginning of the study, at the end of the implementation of the set of preventive interventions, and three months after the end of the implementation.

ELIGIBILITY:
Inclusion Criteria:

* vulnerable elderly 65years and older,
* vulnerable elderly with preserved cognitive abilities,
* vulnerable elderly receiving at least one medication for any medical condition,
* vulnerable elderly treated by a community nurse,
* community-dwelling vulnerable elderly,
* suboptimal adherent vulnerable elderly.

Exclusion Criteria:

* vulnerable elderly with psychoses or dementia,
* vulnerable elderly with cognitive disorders,
* vulnerable elderly addicted to alcohol,
* vulnerable elderly addicted to illegal drugs,
* vulnerable elderly in the terminal phase of the disease (life expectancy less than 6 months).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 639 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in adherence | From date of randomization until final check of changes in adherence and self-efficacy, assessed up to 30 weeks.
  Medication adherence will be assessed using the Tool of adherence behavior screening (TABS), which is a part of the Beliefs and Behavior Questionnaire (BBQ) (George, et al., 2006) and is intended to assess adherence and related behaviors, health beliefs, and experiences of patients with chronic diseases.
  The TABS is a tool that measures patient self-reported adherence (George, et al., 2006). It has two subscales - 'adherence' (statements 2, 3, 4, 5) and 'non-adherence' (statements 1, 6, 7 and 8). Each one contains four statements, to which the respondent decides on a 5-point Likert scale ('never' - 1 to 'always' - 5). We add the points of both subscales and subtract the sum of the points of the subscale 'non-adherence' from the sum of the points of the subscale 'adherence'. In good adherence, the difference is ≥ 15 and in the case of suboptimal adherence, the difference is ≤ 14 (George, et al., 2006).
Change in self-efficacy | From date of randomization until final check of changes in adherence and self-efficacy, assessed up to 30 weeks.
  Self-efficacy will be measured using Self-Efficacy for Appropriate Medication Use (SEAMS) consisting of 13 statements/questions and a 3-point Likert scale (Risser, et al., 2007). The higher the number of points collected, the better the self-efficacy (Risser et al., 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Martina Horvat, Principal Investigator — University of Maribor, Faculty of Health Sciences
Locations (1):
- University of Maribor, Faculty of Health Sciences, Maribor, Styria, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George J, Mackinnon A, Kong DC, Stewart K. Development and validation of the Beliefs and Behaviour Questionnaire (BBQ). Patient Educ Couns. 2006 Dec;64(1-3):50-60. doi: 10.1016/j.pec.2005.11.010. Epub 2006 Jul 14. PMID 16843634
- [Background] Risser J, Jacobson TA, Kripalani S. Development and psychometric evaluation of the Self-efficacy for Appropriate Medication Use Scale (SEAMS) in low-literacy patients with chronic disease. J Nurs Meas. 2007;15(3):203-19. doi: 10.1891/106137407783095757. PMID 18232619